CLINICAL TRIAL: NCT07070622
Title: Planed Organ Preservation for Early- and Intermediate-risk Low Rectal Cancer With Good Response to Neoadjuvant Chemotherapy
Brief Title: Planed Organ Preservation for Low Rectal Cancer After Neoadjuvant Chemotherapy (OPLAR)
Acronym: OPLAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPLAR
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNT (Experimental): During concurrent radiotherapy, capecitabine (825mg/m2, bid, 5d/w) and oxaliplatin (130mg/m2, d1, q3w) were given for 2 cycles. After radiotherapy, two cycles of XELOX chemotherapy were given, with the specific doses of oxaliplatin 130mg/m2, d1, capecitabine 1000mg/m2, D1-14, q3w. Intensity-modulated radiotherapy (IMRT/VMAT) was used for radiotherapy with a dose of 50-50.4Gy/25-28f, 1.8-2.0Gy/d, 5f/w.
  Interventions: Drug: patients were assigned to receive TNT or iTNT management
- iTNT (Experimental): Long-term radiotherapy concurrent with oxaliplatin/capecitabine chemotherapy + tillizumab immunotherapy, concurrent radiotherapy with capecitabine: 825mg/m2, bid, 5d/w, oxaliplatin: 130mg/m2, d1, q3w, tillizumab: 200mg, q3w, 2 cycles. After radiotherapy, two cycles of XELOX+ tislelizumab were given, with the specific doses of oxaliplatin 130mg/m2, d1, capecitabine 1000mg/m2, D1-14, q3w, and tislelizumab 200mg, q3w. Intensity-modulated radiotherapy (IMRT/VMAT) was used for radiotherapy with a dose of 50-50.4Gy/25-28f, 1.8-2.0Gy/d, 5f/w.
  Interventions: Drug: patients were assigned to receive TNT or iTNT management

INTERVENTIONS:
Drug: patients were assigned to receive TNT or iTNT management — TNT or iTNT

SUMMARY:
On the basis of our previous study, this project further explored whether patients with effective neoadjuvant chemotherapy can obtain a higher organ preservation rate after total neoadjuvant therapy. This study was designed to enroll patients with low and intermediate-risk rectal cancer. After 2 cycles of XELOX chemotherapy, patients with effective chemotherapy as judged by high-definition MRI of the rectum (the long diameter of the tumor was shortened by ≥30% compared with that before treatment) were randomly divided into two groups. One group was long-course chemoradiotherapy combined with consolidation chemotherapy (TNT group). In the other group, long-term chemoradiotherapy combined with immunotherapy and consolidation chemotherapy (iTNT group), we explored whether TNT could achieve a higher organ preservation rate after effective neoadjuvant chemotherapy in patients with low and intermediate-risk low rectal cancer, and the organ preservation rate of TNT combined with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old; Gender is not limited;
2. rectal adenocarcinoma confirmed by pathology and pMMR/MSS by immunohistochemistry and/or genetic testing;
3. The following characteristics of the tumor were evaluated by thoracoabdominal CT, rectal ultrasound and MRI: ① The distance between the lower edge of the tumor and the anal verge was ≤5cm measured by digital rectal examination or MRI; ② Clinical stage cT1-3abN0-1M0 (if cT1N0, patients suitable for endoscopic resection should be excluded); ③MRF (-) (> 1mm), EMVI (±); ④ Lateral lymph nodes were negative and less than 7mm; ⑤ tumor diameter ≤5cm; ⑥ tumor circumference ≤2/3.
4. ECOG score: 0-1;
5. Patients with primary rectal cancer did not receive surgery, radiotherapy, chemotherapy or other anti-tumor treatment before enrollment;
6. Normal main organ function, which met the following characteristics: ① Blood routine examination criteria: HB ≥9g/dL, WBC ≥ 3.5/4.0×109/L, neutrophil ≥ 1.5×109/L, PLT≥ 100×109/L; ② Biochemical examination should meet the following criteria: Crea and BIL ≤ 1.0 times the upper limit of normal value (ULN), ALT and AST≤ 2.5 times the upper limit of normal value (ULN), alkaline phosphatase (ALP) ≤2.5×UNL, total bilirubin (Tbil) ≤1.5×UNL.
7. No history of allergy to 5-Fu or platinum drugs; Women of childbearing age were required to have a negative pregnancy test (serum or urine) 7 days before enrollment and to be willing to use an appropriate method of contraception during the trial and for 8 weeks after the last dose. For men, surgical sterilization or consent to use an appropriate method of contraception for the duration of the trial or for 8 weeks after the last dose;

(9) The subjects voluntarily joined the study, signed the informed consent form, with good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. patients with lynch syndrome;
2. Distant metastasis was not considered at initial diagnosis but proved during treatment;
3. previous or concurrent history of other malignant tumors (including synchronous colon cancer), except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
4. patients who had received pelvic radiotherapy;
5. pregnant or lactating women with fertility needs; Male patients with fertility needs;
6. The presence of uncontrolled systemic diseases as determined by the investigator, including diabetes mellitus, hypertension, active autoimmune diseases or a history of autoimmune diseases (e.g., interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism), and severe heart, lung, and kidney diseases; Subjects had active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL) and hepatitis C (hepatitis C antibody positive and HCV-RNA higher than the detection limit of the analytical method).
7. those with mental disorders;
8. Severe infection (CTCAE > 2) occurred within 4 weeks before the first dose of study drug, such as severe pneumonia requiring hospitalization, bacteremia, and infectious complications; Patients with active pulmonary inflammation on baseline chest imaging or signs and symptoms of infection requiring treatment with oral or intravenous antibiotics within 2 weeks before the first dose of study drug were excluded if prophylactic antibiotics were used.
9. patients with bleeding diathesis or coagulopathy were on thrombolytic/anticoagulant therapy; Aneurysm, stroke, transient ischemic attack, arteriovenous malformation in the past year;
10. serious gastrointestinal diseases affecting the absorption of oral chemotherapy drugs, and a history of gastrointestinal fistula, perforation, bleeding or severe ulcer;
11. a history of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplantation or allogeneic bone marrow transplantation;
12. patients with a history of interstitial lung disease, noninfectious pneumonia, pulmonary fibrosis or other uncontrolled acute lung disease, active pulmonary tuberculosis infection detected by medical history or CT examination, or a history of active pulmonary tuberculosis infection within 1 year before enrollment, or a history of active pulmonary tuberculosis infection more than 1 year before enrollment but without regular treatment;
13. known allergic to macromolecular protein preparations, or to any component of tislelizumab, or allergic, hypersensitive, or contraindicated to etoposide or cisplatin or any component used in their preparations;
14. have received or are receiving any of the following therapies: a. Anti-pd-1 or anti-PD-L1 antibody therapy, chemotherapy, radiotherapy, targeted therapy; b. received any study drug within 4 weeks before the first dose of the study drug; c. subjects requiring systemic treatment with corticosteroids (> 10 mg prednisone equivalent daily) or other immunosuppressive agents within 2 weeks before the first dose of study drug, except when corticosteroids are used for local inflammation and to prevent allergy, nausea, and vomiting. Other special circumstances require communication with the sponsor. In the absence of active autoimmune disease, inhaled or topical steroids and adrenocortical hormone replacement at a therapeutic dose of prednisone of more than 10mg per day were allowed. d. vaccination with an antitumor vaccine or live vaccine within 4 weeks before the first dose of study drug;
15. enrolled in an additional clinical trial within 4 weeks before initiation of treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
organ preservation rate，OPR | no recurrence within 2 years
  ① The number of patients with cCR or near cCR at 8 weeks after radiotherapy who chose watchful waiting and sustained cCR for 2 years;
  ② Patients were evaluated as cCR or near cCR at 8 weeks after the end of radiotherapy, entered watchful waiting, and finally selected local resection, and there was no recurrence within 2 years after local resection, and no additional salvage surgery.

SECONDARY OUTCOMES:
DFS | 3 years
  disease free survival
OS | 3 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No